CLINICAL TRIAL: NCT05912634
Title: Early Complication and Outcomes in Surgical vs no Surgical Involvement of Aortic Arch in Type A Aortic Dissection
Brief Title: Repair Versus Non-repair of the Aortic Arch in Type A Aortic Dissection
Acronym: AoArch
Status: Enrolling by invitation | Type: Observational
Sponsor: Centre Cardiologique du Nord (Other)
Collaborators: Henri Mondor University Hospital (Other); Universita degli Studi di Genova (Other); Pitié-Salpêtrière Hospital (Other)
Responsible Party: Principal Investigator, Francesco Nappi, Director, Centre Cardiologique du Nord
Other Study IDs: CN-202201173-2; CN-23-27 (Other: Centre Cardiologique du Nord)
Record Dates: First submitted 2023-05-30; First posted 2023-06-22 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Aortic Dissection; Aortic Arch; Aortic Dissection Rupture; Aortic Dilatation
Keywords: Type A Aortic Dissection (TAAAD); Root-Sparing Replacement; Ascending Aorta Replacement; Partial Arch Repair; Total Arch Replacement (TARP); Frozen Elephant Trunk (FET); Hemiarch Procedures
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conservative Type A Aortic Dissection Repair (TAAD-R): The Conservative procedure will include patients receiving ascending aortic root sparing replacement with or without the implantation of the aortic hemiarch
  Interventions: Procedure: Conservative TAAD-R
- Extensive Type A Acute Aortic Dissection Repair (TAAD-R): The extensive procedure will include patients receiving ascending aorta replacement associated to TARP
  Interventions: Procedure: Extensive TAAD- R

INTERVENTIONS:
Procedure: Conservative TAAD-R — Cardiac arrest will be ensured using antegrade potassium-rich cardioplegia solution delivered directly into the coronary ostium or after coronary sinus cannula insertion, in patients with aortic regurgitation aorta will be resected down to the sinotubular junction and the thrombus located in the false lumen of the aortic root will be removed so that the aortic lesion could be visualized. The commissures will be resuspended using 4-0 or 5-0 sutures reinforced with a Teflon pledget over each commissure. A 4-0 or 5-0 polypropylene suture will be chosen to seal the proximal anastomosis and this suture line will also be used to secure the intima to the adventitia. In patients revealing normal-sized aortic roots associated with poor-quality valve leaflets, concomitant aortic valve replacement with conventional xenograft or mechanical prosthesis will be preferred.
  Other Names: Ascending Aortic Root Sparing Replacement with or without Hemiarch Repair
  Groups: Conservative Type A Aortic Dissection Repair (TAAD-R)
Procedure: Extensive TAAD- R — Patients who experienced dilatation of the sinuses of Valsalva >4.5 cm in diameter on computed tomography imaging, those with connective tissue disease, or those in whom intimal tears extended into the sinuses, will undergoing replacement of the aortic root using a biologic or mechanical composite valve graft or valve-sparing root reimplantation procedure.Total arch replacement procedures (TARP) will fulfilled with the use of deep hypothermic circulatory arrest and with either antegrade or retrograde cerebral perfusion, maintaining systemic cooling between 19°C to 25°C and depending on the surgeon's practice.TARPs will be carried out using 1- and 4-branch grafts and involved the resection of all the aortic tissue up to the left common carotid artery (total arch)
  Other Names: Aortic root procedures.TARP procedures. Frozen Elephant Trunk (FET) procedure
  Groups: Extensive Type A Acute Aortic Dissection Repair (TAAD-R)

SUMMARY:
Acute Stanford type A aortic dissection (TAAD) is a life-threatening clinical status requiring surgery that is usually performed as a salvage procedure.We planned a multicenter study to evaluate the balance between the patient's condition and those therapeutic strategies that may limit the risk of late adverse events in patients who will be underwent surgery for appropriate management of TAAD

DETAILED DESCRIPTION:
Substantial evidence has suggested a decrease of early mortality during the last years, however recently the Nordic Consortium for Acute Type A Aortic Dissection registry recorded 18% of 30-day mortality after surgery for ATAAD. Similarly, the prospective German Registry for Acute Aortic Dissection Type A confirmed this data reporting a 30-day mortality of 16.9%. Again, results from recent analysis of the Society of Thoracic Surgeon database that report 7353 procedures from 2014 and 2017 for acute TAAD revealed a 30-day mortality of 17%. Understanding the balance between the patient's conditions which may not allow extensive procedure and those treatment strategies which may limit the risk of late adverse events in patients who remain alive long after the surgery is essential for an appropriate management of ATAAD. The best treatment option in patients with ATAAD is dictated by the balance between patient conditions that may not allow for extensive procedures and those more conservative treatment strategies that limit the risk of late adverse events in patients who remain alive long after surgery. surgery. However, previous evidence from large series of patients do not provide information on the long-term durability of these procedures.

Here investigators planned a multicenter study to evaluate the contemporary early outcomes and duration of different surgical strategies for 15-year acute ATAAD in a large study population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years
* TAAD or intramural hematoma involving the ascending aorta
* Symptoms started within 7 days from surgery
* Primary surgical repair of acute TAAD
* Any other major cardiac surgical procedure concomitant with surgery for TAAD.

Exclusion Criteria:

* Patients aged < 18 years
* Onset of symptoms > 7 days from surgery
* Prior procedure for TAAD
* Concomitant endocarditis;
* TAAD secondary to blunt or penetrating chest trauma.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The retrospective multicenter study including patients who underwent surgery for acute TAAAD at 5 centers of cardiac surgery located in 2 European countries and Japan (2 France, 2 Italy and 1 Hokkaido ). Data will be prospectively collected fron patients (conservative vs estensive TAAD- R) treated during the study period and the aim will be to gather further data for future clinical research on this topic. Preoperative and postoperative variables will be included during in-hospital stay and follow-up data instead they will be included on subsequent encounters for all other patients who will be hospitalized. Data on consecutive patients with acute TAAD will be collected with pre-specified baseline, operative and outcome variables.
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Operative Mortality (OM) | 30-day
  Patients who died within 30 days
Rate of acute heart failure | 30-day
  Number of participants with postoperative heart failure who will require prolonged use of concentration of inotropes for a period greater than 24 h and/or the insertion of any mechanical circulatory support device.
Stroke | 30-day
  Number of participants with acute episode of a focal or global neurological deficit. Rates of alteration of degree of consciousness, hemiplegia, hemiparesis, numbness or sensory loss affecting one side of the body, dysphasia or aphasia, hemianopsia, amaurosis fugax. To consider rate of other neurologic signs or symptoms consistent with stroke duration of focal or global neurologic deficit greater than 24 hours.
Rate of global brain ischemia | 30-days
  Rate of diffuse hypoxic damage as diagnosed at brain imaging and electroencephalography.
Rate of mesenteric ischemia | 30-days
  Rate of abdominal pain with or without nausea and vomiting and rectal bleeding or bloody diarrhea
Rate of acute kidney injury | 30-days
  Number of participants with postoperative change in serum creatinine concentration. Severity will be stratified on the basis of number of participants with the KDIGO (Kney Disease Improving Global Outcomes) criteria.

SECONDARY OUTCOMES:
Rate of paraplegia/paraparesis | 30-day
  Rate of bilateral weakness and/or multimodality sensory disturb- ance below the level of the ischemic spinal lesion.
Rate of perioperative bleeding | 30-day
  Number of participants will receive postoprative transfused red blood cell units. The E-CABG ( coronary artery by pass grafting) classification of bleeding rate has been proposed as a simple classification of perioperative bleeding
Rate of reoperation for bleeding | 30-day
  Number of participants who will receive postoperative chest reopening for excessive bleeding.
Rate of mechanical circulatory support | 30-day
  Number of participants who will receive the use of intra-aortic balloon pump and/or venoarterial extracorporeal membrane oxygenation for postoperative acute heart failure.
Late outcomes | 18 years
  Data on patient's survival status will be collected

OTHER OUTCOMES:
Rate of urgent procedure | 30-days
  Number of participants who will require scheduled procedure within 24 hours of admission.
Rate of emergency grade 1 | 30-days
  Number of participants will require procedure within 24 hours of hospital admission and who are symptomatic or minimally symptomatic with stable hemodynamic conditions and no signs of malperfusion.
Rate of emergency grade 2 | 30-days
  Number of participants who will require procedure within the first 6 hours of hospital admission due to hemodynamic instability despite use of concentration inotropes and/or malperfusion.
Rate of salvage grade 1 | 30-days
  Number of participants who will require immediate surgical procedure. Rate of cardio pulmonary resuscitation with external chest compressions and/or open cardiac massage between induction of anesthesia and initiation of cardiopulmonary bypass.
Rate of salvage grade 2 | 30-days
  Number of participants who will require immediate surgical procedure. Rate of cardiopulmonary resuscitation with external chest compressions en route to the operating theatre or prior to induction of anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Nappi, Study Chair — Cardiac Surgery Centre Cardiologique du Nord de Saint-Denis, Paris, France
Locations (1):
- Francesco Nappi, Saint-Denis, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Geirsson A, Shioda K, Olsson C, Ahlsson A, Gunn J, Hansson EC, Hjortdal V, Jeppsson A, Mennander A, Wickbom A, Zindovic I, Gudbjartsson T. Differential outcomes of open and clamp-on distal anastomosis techniques in acute type A aortic dissection. J Thorac Cardiovasc Surg. 2019 May;157(5):1750-1758. doi: 10.1016/j.jtcvs.2018.09.020. Epub 2018 Sep 29. PMID 30401530
- [Result] Harris KM, Nienaber CA, Peterson MD, Woznicki EM, Braverman AC, Trimarchi S, Myrmel T, Pyeritz R, Hutchison S, Strauss C, Ehrlich MP, Gleason TG, Korach A, Montgomery DG, Isselbacher EM, Eagle KA. Early Mortality in Type A Acute Aortic Dissection: Insights From the International Registry of Acute Aortic Dissection. JAMA Cardiol. 2022 Oct 1;7(10):1009-1015. doi: 10.1001/jamacardio.2022.2718. PMID 36001309
- [Result] Benedetto U, Dimagli A, Kaura A, Sinha S, Mariscalco G, Krasopoulos G, Moorjani N, Field M, Uday T, Kendal S, Cooper G, Uppal R, Bilal H, Mascaro J, Goodwin A, Angelini G, Tsang G, Akowuah E. Determinants of outcomes following surgery for type A acute aortic dissection: the UK National Adult Cardiac Surgical Audit. Eur Heart J. 2021 Dec 28;43(1):44-52. doi: 10.1093/eurheartj/ehab586. PMID 34468733
- [Result] O'Hara D, McLarty A, Sun E, Itagaki S, Tannous H, Chu D, Egorova N, Chikwe J. Type-A Aortic Dissection and Cerebral Perfusion: The Society of Thoracic Surgeons Database Analysis. Ann Thorac Surg. 2020 Nov;110(5):1461-1467. doi: 10.1016/j.athoracsur.2020.04.144. Epub 2020 Jun 26. PMID 32599034
- [Result] Czerny M, Schoenhoff F, Etz C, Englberger L, Khaladj N, Zierer A, Weigang E, Hoffmann I, Blettner M, Carrel TP. The Impact of Pre-Operative Malperfusion on Outcome in Acute Type A Aortic Dissection: Results From the GERAADA Registry. J Am Coll Cardiol. 2015 Jun 23;65(24):2628-2635. doi: 10.1016/j.jacc.2015.04.030. PMID 26088302